CLINICAL TRIAL: NCT04368533
Title: A Pilot Study to Evaluate the Effect of Livionex on Reducing Plaque Accumulation and Improving Oral Health in Children
Brief Title: Livionex on Reducing Plaque Accumulation and Improving Oral Health in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 17-22447
Record Dates: First submitted 2019-01-25; First posted 2020-04-29 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Plaque, Dental; Caries, Dental; Oral Hygiene
Keywords: Livionex dental gel, toothpaste
MeSH Terms: conditions — Dental Plaque; Dental Caries

STUDY DESIGN:
Intervention Model Description: double-blind randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Livionex Dental Gel (Experimental): Children assigned to this arm will brush/clean teeth with Livionex Dental Gel twice a day for up to 12 months.They will undergo a dental exam by a trained dentist including caries assessment (at baseline, 1, 3, 6, 9 or 12 months), dental plaque photograph, (at baseline, 1, 3, 6 and 9 or 12 months), and swab samples for dental plaque and saliva will be collected at all study visits. A questionnaire will be given to address dentifrice and brushing experience. Data on compliance and side-effects of toothpastes will be collected at each of the calls.
  Interventions: Drug: Livionex Dental Gel
- A standard children's toothpaste containing 1500 ppm fluoride (Active Comparator): Children assigned to this arm will brush/clean teeth with a standard children's toothpaste containing 1500 ppm fluoride twice a day for up to 12 months. They will undergo a dental exam by a trained dentist including caries assessment (at baseline, 1, 3, 6, 9 or 12 months), dental plaque photograph, (at baseline, 1, 3, 6, 9 or 12 months), and swab samples for dental plaque and saliva will be collected at all study visits. A questionnaire will be given to address dentifrice and brushing experience at each study visit. A monthly phone call will be made to assess compliance with the study protocol, and to answer any questions or concerns. Data on compliance and side-effects of toothpastes will be collected at each of the calls.
  Interventions: Drug: A standard children's toothpaste containing 1500 ppm fluoride

INTERVENTIONS:
Drug: Livionex Dental Gel — The subjects will brush their teeth with Livionex Dental Gel twice a day for up to 12 months.
  Arms: Livionex Dental Gel
Drug: A standard children's toothpaste containing 1500 ppm fluoride — The subjects will brush their teeth with a standard children's toothpaste containing 1500 ppm fluoride twice a day for up to 12 months.
  Arms: A standard children's toothpaste containing 1500 ppm fluoride

SUMMARY:
This is an investigator initiated randomized double-blind pilot study at the UCSF Pediatric Dental Clinics to compare effectiveness of a new toothpaste Livionex Dental Gel with a standard children's toothpaste containing 1500 ppm fluoride in reducing dental plaque and caries in healthy and well children every 3 months for up to 12 months.

DETAILED DESCRIPTION:
Dental plaque is the primary etiological factor in the initiation of caries, gingival inflammation and subsequent destruction of periodontal tissues. Effective oral hygiene eliminates microbial plaque leading to resolution of gingival inflammation. Livionex Dental Gel is a toothpaste that is effective in reducing plaque in adults while not containing the additives found in other toothpastes that can cause increased gingival irritation. The investigators hypothesize that brushing with Livionex toothpaste creates an oral environment that prevents dental plaque accumulation and promotes oral health in children.

This study will prospectively enroll 78 children aged 9 months to 12 years from UCSF pediatric dental clinics. Upon obtaining an informed consent, children will be randomized in a 1:1 ratio to the use of test (Livionex Dental Gel) and control toothpaste (a standard children's toothpaste containing 1500 ppm fluoride ). All patients will be provided a soft brush at enrollment, and the child and/or the parent will be taught to brush/clean after the first exam, with the assigned dentifrice, at the study center before they go home. Additionally, each subject will receive a new brush at every 3-month visit. Subjects will undergo a dental exam by a trained dentist including caries assessment (at baseline, 1, 3, 6, 9 or 12 months), dental plaque photograph, (at baseline, 1, 3, 6 and 9 or 12 months), and swab samples for dental plaque and saliva will be collected at all study visits. A questionnaire will be given to address dentifrice and brushing experience in a phone call one month after enrollment and at the last study visit. Data on compliance and side effects of toothpastes will be collected at each of the calls.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 9 months to 12 years.
* Parent and children are able complete the study procedures.
* Parent/legal guardian willing to allow their child participate and sign informed consent form.

Exclusion Criteria:

* Parents are unable to understand or participate in study procedures.
* Known allergy to edathamil or known allergy to multiple hygiene and cosmetic products.

Ages: 9 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Changes of dental plaque | up to 12 months
  To compare plaque reduction between Livionex Dental Gel and control toothpaste group from baseline to 1, 3, 6 and 9/12 months months. Plaque will be assessed using a plaque index score (Turesky modification of the Quigley-Hein Plaque Index) for each tooth and a total plaque score will be divided by the number of teeth present for analysis.
Incidence of new dental caries. | up to 12 months
  To compare incidence of new dental caries between Livionex Dental Gel and control toothpaste group from baseline to 1, 3, 6 and 9/12 months.
Changes of oral microbiome composition | up to 12 months
  Using 16S rRNA gene sequences and taxonomic annotation to identify dental caries relevant pathogenic, commensal, and probiotic bacteria and archaea and to compare temporal changes in oral microbiome composition, diversity and relative quantity between Livionex Dental Gel and control toothpaste group from baseline to 1, 3, 6 and 9/12 months months.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Den-Besten, DDS, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Pediatric Dentistry Parnassus Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dadkhah M, Chung NE, Ajdaharian J, Wink C, Klokkevold P, Wilder-Smith P. Effects of a Novel Dental Gel on Plaque and Gingivitis: A Comparative Study. Dentistry (Sunnyvale). 2014 Jun 1;4(6):239. doi: 10.4172/2161-1122.1000239. PMID 26052472
- [Background] Bowen WH, Koo H. Biology of Streptococcus mutans-derived glucosyltransferases: role in extracellular matrix formation of cariogenic biofilms. Caries Res. 2011;45(1):69-86. doi: 10.1159/000324598. Epub 2011 Feb 23. PMID 21346355
- [Background] Raad II, Fang X, Keutgen XM, Jiang Y, Sherertz R, Hachem R. The role of chelators in preventing biofilm formation and catheter-related bloodstream infections. Curr Opin Infect Dis. 2008 Aug;21(4):385-92. doi: 10.1097/QCO.0b013e32830634d8. PMID 18594291
- [Background] Pitts NB, Ekstrand KR; ICDAS Foundation. International Caries Detection and Assessment System (ICDAS) and its International Caries Classification and Management System (ICCMS) - methods for staging of the caries process and enabling dentists to manage caries. Community Dent Oral Epidemiol. 2013 Feb;41(1):e41-52. doi: 10.1111/cdoe.12025. PMID 24916677
- [Background] Soderling E, Isokangas P, Pienihakkinen K, Tenovuo J. Influence of maternal xylitol consumption on acquisition of mutans streptococci by infants. J Dent Res. 2000 Mar;79(3):882-7. doi: 10.1177/00220345000790031601. PMID 10765964
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] van der Weijden GA, Hioe KP. A systematic review of the effectiveness of self-performed mechanical plaque removal in adults with gingivitis using a manual toothbrush. J Clin Periodontol. 2005;32 Suppl 6:214-28. doi: 10.1111/j.1600-051X.2005.00795.x. PMID 16128840
- [Background] Wu H, Moser C, Wang HZ, Hoiby N, Song ZJ. Strategies for combating bacterial biofilm infections. Int J Oral Sci. 2015 Mar 23;7(1):1-7. doi: 10.1038/ijos.2014.65. PMID 25504208
- [Background] Young DA, Featherstone JD. Caries management by risk assessment. Community Dent Oral Epidemiol. 2013 Feb;41(1):e53-63. doi: 10.1111/cdoe.12031. PMID 24916678
- [Background] Zhan L, Cheng J, Chang P, Ngo M, Denbesten PK, Hoover CI, Featherstone JD. Effects of xylitol wipes on cariogenic bacteria and caries in young children. J Dent Res. 2012 Jul;91(7 Suppl):85S-90S. doi: 10.1177/0022034511434354. PMID 22699675